CLINICAL TRIAL: NCT03505086
Title: Bleeding in Thrombocytopenia Explained
Acronym: BITE
Status: Recruiting | Type: Observational
Sponsor: Sanquin-LUMC J.J van Rood Center for Clinical Transfusion Research (Other)
Responsible Party: Sponsor
Other Study IDs: PPOC 17-36
Record Dates: First submitted 2018-02-06; First posted 2018-04-23 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Hematologic Neoplasms; Bleeding; Hemorrhage; Platelet Transfusion
MeSH Terms: conditions — Hematologic Neoplasms; Hemorrhage | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Citrate plasma and urine. NB: not all enrolled patients will be elligible for sampling, some enrolled patients are only elligible for epidemiological study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cohort: All patients fulfilling the eligibility criteria who can be asked for consent. Basic register of only patient diagnosis, treatment and bleeding yes or no (without identifiable information).
- cases: Patient with clinically relevant bleeding, defined as major and clinically relevant non-major bleeding that leads to substantial additional medical care: WHO score 3-4 and part of the WHO score 2 bleedings (depending on the need for additional care).
  Interventions: Diagnostic Test: Blood withdrawal; Other: Questionnaire for former bleeding events
- controls: Patient without clinically relevant bleeding matched to a case patient based on diagnosis and therapy.
  Interventions: Diagnostic Test: Blood withdrawal; Other: Questionnaire for former bleeding events

INTERVENTIONS:
Diagnostic Test: Blood withdrawal — * Blood withdrawal will be at regular sampling moments, blood can be collected from a central venous catheter or venepuncture procedure.
  * Blood withdrawal will be performed for a maximum of 10 times per admission, 10 ml per time.
  * Urine sampling will be for a maximum of 5 times per admission.
  * Urine can be sampled from a catheter when present, or collected regular.
  Other Names: Collection of urine (with or without catheter)
  Groups: cases; controls
Other: Questionnaire for former bleeding events — Questionnaire to investigate a bleeding tendency before diagnosis.
  Groups: cases; controls

SUMMARY:
Multicenter case cohort study investigating clinical risk factors for clinically relevant bleeding in hemato-oncology patients, as well as bleeding related biomarkers during intensive treatment.

DETAILED DESCRIPTION:
Rationale: Hemato-oncological patients treated with intensive chemotherapy receive prophylactic platelet transfusions to prevent bleeding events as soon as their platelet counts drop below 10 x109/L. This platelet count based prophylactic transfusion strategy, however, is both inefficient and often not needed. This is reflected in the high percentage of patients with bleeding despite this strategy (43%), and the high percentage of patients who do not bleed without this strategy (50%). Solely platelet count therefore is not a good predictor for bleeding. Identification of new risk factors and confirmation of already suspected risk factors is essential, and should lead to better prediction and prevention of bleeding. Patients with a high risk profile could be given more effective haemostatic treatments including more efficient transfusion strategies. On the other hand one could consider omitting prophylactic transfusions to low risk patients and conditions. Furthermore, additional knowledge about the pathophysiology of bleeding in hemato-oncology patients is needed.

Objective: Identify hemato-oncology patients and conditions with a high versus a low bleeding risk and investigate the association of bleeding related biomarkers with bleeding.

Study design: Case cohort study, consisting of two parts: epidemiologically research including short questionnaire (part A, eligible for all patients fulfilling inclusion criteria), and additional blood and urine sampling (part B, eligible only for included patients admitted for chemotherapy or stem cell transplantation).

Study population: Adult hemato-oncology patients: 1.) who are admitted for treatment and who have or will develop thrombocytopenia and are likely to receive one or more prophylactic platelet transfusions, and 2.) patients who have received such treatments in the last year but are readmitted to the hospital for disease or treatment related adverse events.

Intervention: Part A: standard available data collection, short questionnaire. Part B: sampling of blood and urine on top of routinely performed laboratory tests.

Main study parameters: Part A: The presence of clinical factors and results of routinely performed laboratory tests compared between bleeding versus non-bleeding patients. Part B: Presence of markers for coagulation-, platelet- and endothelial or vascular dysfunction compared between bleeding versus non-bleeding patients.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Part A: No burden or health risks: comparison of standard available data between bleeding and non-bleeding patients makes this a non-WMO part of the study, since there is no invasive intervention. The 10-15 minutes questionnaire in this respect is not considered as a burden. Part B of the study only applies for a subgroup of the included patients and falls under the scope of the WMO. The intervention is the additional to regularly performed citrate anticoagulated blood sampling (maximum 10 samples of 10-15 cc in 4 weeks), as well as weekly urine sampling. Both are considered a minor burden for participants, and the risk of additional blood sampling at regular sampling moments is negligible. Finally, all BITE-study activities in both study parts will not have any consequences on the treatment or monitoring of patients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are mentioned below and differ for part A and B of the study.

* Admission in the hospital. (part A and B)
* Age ≥ 18 years. (part A and B)

AND:

• Hemato-oncology patient, including MDS and AA, admitted for treatment (chemotherapy, SCT) who is (expected to become) thrombocytopenic with platelet counts of < 50 for expected at least 5 days and who will possibly be treated with one or more prophylactic platelet transfusions. (part A and B)

OR:

• Hemato-oncology patient who had previous intensive chemotherapy or stem cell transplantation and who is admitted to the hematology ward for disease or treatment related events or complications. (part A only)

Exclusion Criteria:

• Patients with myeloproliferative disorders.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hemato-oncology patients
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinically relevant bleeding events | Bleeding must occur during hospital admission, which on average will be 3-4 weeks.
  Bleeding events that are clinically relevant. i.e. all WHO grade 3 and 4 bleedings, as well as WHO grade 2 bleedings that lead to substantial additional medical care (ISTH criteria).
  We will quantify the association of possible risk factors for bleeding with this primary outcome. These risk factors are listed in the protocol.

SECONDARY OUTCOMES:
Mortality | During hospital admission, which on average will be 3-4 weeks.
  Mortality during hospital stay in bleeding vs non-bleeding patients
Duration of hospital stay | At the day of discharge, which will be on average 3-4 weeks.
  Duration of hospital stay in bleeding vs non-bleeding patients

CONTACTS AND LOCATIONS:
Locations (1):
- LUMC, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cornelissen LL, Caram-Deelder C, van der Bom JG, Middelburg RA, Zwaginga JJ. Risk factors for bleeding in haemato-oncology patients-a nested case-control study: The BITE study protocol (Bleeding In Thrombocytopenia Explained). BMJ Open. 2020 Jun 30;10(6):e034710. doi: 10.1136/bmjopen-2019-034710. PMID 32606056